CLINICAL TRIAL: NCT07067489
Title: The Effect of Whole-Body Vibration Exercises Combined With Balneotherapy on Pain, Function, and Sleep Quality in Patients With Chronic Low Back Pain
Brief Title: Whole-Body Vibration and Balneotherapy in Chronic Low Back Pain
Acronym: Whole-Body Vib
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Selim Mahmut GÜNAY, Asst prof, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025/8-3
Record Dates: First submitted 2025-07-03; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Balneology; Whole Body Vibration; Water; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Balneology

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balneotherapy and Standard Exercise Group (Experimental): Participants in this group will receive 20-minute balneotherapy sessions five days per week for three weeks. Following a 30-40 minute rest, they will perform a standardized exercise program targeting chronic low back pain. The program includes stretching, strengthening, range of motion, and stabilization exercises focused on the lumbar spine, hips, and lower extremities. Exercises will be performed in 2 sets of 8-10 repetitions. Sessions will be supervised by a physiotherapist.
  Interventions: Behavioral: Balneotherapy
- Balneotherapy and Whole-Body Vibration Exercise Group (Experimental): Participants in this group will also receive 20-minute balneotherapy sessions five days per week for three weeks. After a 30-40 minute rest, they will first complete the same standardized exercise program as the first group. Then, they will perform whole-body vibration (WBV) exercises on a vibration platform (Compex Winplate). The WBV session will include static squats, dynamic squats, bridge exercises, dynamic weight shifting, and toe raises, performed at 30-40 Hz frequency and 2-4 mm amplitude for 40-60 seconds per set, with 2 sets per session and 3-minute rest intervals.
  Interventions: Behavioral: Balneotherapy; Behavioral: Whole-Body Vibration Exercise

INTERVENTIONS:
Behavioral: Balneotherapy — Participants receive 20-minute balneotherapy sessions involving full-body immersion in thermal-mineral spring water at a therapeutic spa facility. Sessions are conducted five days per week over a three-week period. Water temperature and mineral content are standardized according to institutional protocols. The intervention is designed to provide analgesic, anti-inflammatory, and muscle-relaxant effects through thermally induced vasodilation and neuromuscular modulation.
Behavioral: Whole-Body Vibration Exercise — Participants perform whole-body vibration (WBV) exercises using the "Compex Winplate" platform (Uniphy Elektromedizin GmbH & CoKG), certified under ISO 9001:2000 and DIN EN ISO 13485:2003. The exercise protocol includes static squats, dynamic squats, bridge exercises, dynamic weight shifting, and toe raises. Vibration is applied at a frequency of 30-40 Hz and amplitude of 2-4 mm for 40-60 seconds per set, with two sets per session and a 3-minute rest between sets. WBV is applied following a standardized exercise program, and the full intervention is delivered five days per week for three weeks.
  Arms: Balneotherapy and Whole-Body Vibration Exercise Group

SUMMARY:
This randomized controlled clinical trial aims to investigate the effects of whole-body vibration (WBV) exercises combined with balneotherapy on pain, physical function, sleep quality, and daily activity levels in individuals with chronic low back pain.

A total of 60 volunteers aged 18 to 65 who have been diagnosed with chronic low back pain by a physical medicine and rehabilitation specialist and who meet the eligibility criteria will be included. Participants will be randomly assigned to two groups. Both groups will receive balneotherapy five days a week for three weeks. After balneotherapy, the first group will perform standard stretching, strengthening, and aerobic exercises designed for low back pain. The second group will receive the same exercise program in combination with WBV exercises using a vibration platform. WBV sessions will include static and dynamic exercises with specific frequency and amplitude settings.

All participants will be evaluated at baseline and after three weeks using validated measures, including pain intensity (Visual Analog Scale), spinal mobility (Modified Schober Test), balance and reach (Functional Reach Test), physical performance (Sit-to-Stand and Timed Up and Go Tests), disability (Oswestry Disability Index, Roland-Morris Questionnaire), and sleep quality (Pittsburgh Sleep Quality Index).

The study seeks to determine whether combining WBV with balneotherapy can provide additional benefits over standard exercise alone in managing chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary consent to participate in the study
* Age between 18 and 65 years
* Having chronic low back pain lasting at least 3 months or recurring at least 3 times per week
* Diagnosis of chronic low back pain by a physical medicine and rehabilitation specialist
* Normal neurological examination findings (no abnormal lower extremity reflexes or anesthesia)

Exclusion Criteria:

* Presence of radicular pain or radiculopathy
* Spondylolisthesis, spinal stenosis, vertebral infection, or cauda equina syndrome
* Vertebral fracture, axial spondyloarthritis
* History of lumbar spine surgery
* Inflammatory rheumatic disease, psychiatric or neurological disorders
* Uncontrolled hypertension, decompensated organ failure, or malignancy
* Pregnancy or breastfeeding
* Use of systemic steroids in the last 3 months
* Major trauma or surgery within the past 6 months
* Receiving physical therapy or physical modalities within the past 6 months
* Any health condition that prevents participation in balneotherapy or exercise programs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Baseline and after 3 weeks of intervention
  SQI will be used to evaluate subjective sleep quality across 7 components. Higher total scores indicate poorer sleep quality.
Functional disability measured by Oswestry Disability Index | Baseline and after 3 weeks of intervention
Modified Schober Test | Baseline and after 3 weeks
Timed Up and Go (TUG) Test | Baseline and after 3 weeks
30-Second Chair Stand Test | Baseline and after 3 weeks
Functional Reach Test | Baseline and after 3 weeks
Roland-Morris Disability Questionnaire | Baseline and after 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dilekci E, Ozkuk K, Kaki B. The short-term effects of balneotherapy on pain, disability and fatigue in patients with chronic low back pain treated with physical therapy: A randomized controlled trial. Complement Ther Med. 2020 Nov;54:102550. doi: 10.1016/j.ctim.2020.102550. Epub 2020 Sep 4. PMID 33183668
- [Background] Blanco-Gimenez P, Vicente-Mampel J, Gargallo P, Baraja-Vegas L, Bautista IJ, Ros-Bernal F, Barrios C. Clinical relevance of combined treatment with exercise in patients with chronic low back pain: a randomized controlled trial. Sci Rep. 2024 Jul 24;14(1):17042. doi: 10.1038/s41598-024-68192-2. PMID 39048701
- [Background] Remer F, Keilani M, Kull P, Crevenna R. Effects of whole-body vibration therapy on pain, functionality, postural stability, and proprioception in patients with subacute and chronic non-specific low back pain: a systematic review. Wien Med Wochenschr. 2025 Feb;175(1-2):20-40. doi: 10.1007/s10354-023-01026-4. Epub 2023 Nov 24. PMID 37999785